CLINICAL TRIAL: NCT01317342
Title: A Randomized Multicenter Study on the Effects of Hypothermic Oxygenated Perfusion (HOPE) on Human Liver Grafts Before Transplantation
Brief Title: Hypothermic Oxygenated Perfusion (HOPE) of Human Liver Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-0079
Record Dates: First submitted 2011-03-10; First posted 2011-03-17 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Injury
Keywords: liver transplantation; machine liver perfusion; extended criteria liver grafts; donation after cardiac death; hypothermic machine liver perfusion; liver reperfusion injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermic oxygenated perfusion (HOPE) (Active Comparator): Application of HOPE for 1 hour
  Interventions: Device: Hypothermic oxygenated perfusion (HOPE)
- Control group: no intervention (No Intervention): Conventional cold storage (IGL-1)

INTERVENTIONS:
Device: Hypothermic oxygenated perfusion (HOPE) — Application of HOPE for 1 hour, perfusion rate 150-300 ml/min, pressure controlled, perfusion pressure < 3 mm Hg, perfusion route portal vein, recirculating system, perfusion volume 2 L, perfusate Institute George Lopez solution (IGL-1), perfusate temperature 4-6 °C, perfusate oxygenation 150-200 mm Hg
  Arms: Hypothermic oxygenated perfusion (HOPE)

SUMMARY:
The purpose of this study is, in a randomized trial, to test a newly developed machine perfusion technique of human liver allografts before transplantation.

Ischemia-reperfusion injury is universal in organ transplantation and leads to varying degrees of graft dysfunction. Despite this fact, the preservation method in organ transplantation has been left unchanged for many years and remains simple static cold storage. Given the scarce donor supply, an increasing number of so called marginal or extended criteria donor organs have been used for liver transplantation, grafts which were previously rarely considered. In addition, allocation policy has changed in many countries, and livers are currently often distributed by the severity of the recipient's disease. As a result, transplant candidates present sicker, with higher MELD (Model for end stage liver disease) scores, at the time of transplant,and the risk of graft dysfunction or even failure due to reperfusion injury is high after the use of marginal livers in sick recipients.

Machine liver perfusion techniques have been significantly improved during the past decade to decrease reperfusion injury, and a number of promising results show beneficial effects in various animal transplant models by either normothermic or hypothermic oxygenated continuous liver perfusion. These techniques generally require machine liver perfusion immediately after organ procurement. However, continuous perfusion has several drawbacks, including major logistic efforts and risk of organ damage during perfusion and transport.

Our group, therefore, focused on the practicability of machine liver perfusion. We developed an endischemic hypothermic oxygenated perfusion (HOPE) concept through the portal vein only. This technique can be easily applied in the operation room shortly before transplantation of the recipient, thus after organ transport and back table preparation.

Recently, the beneficial effect of a similar approach has been confirmed in human liver grafts by a phase I non randomized trial. These results prove feasibility and safety of an endischemic hypothermic machine perfusion approach and warrant further randomized studies.

DETAILED DESCRIPTION:
The study consists on two groups, a perfusion group and a control group. Patients on the waiting list for liver transplantation with proven written consent will be recruited and randomized during organ procurement. Randomization will be performed by computer (secutrial). Perfusion will be started in the operation room after regular organ procurement, transport and back table preparation. The perfusion procedure will not delay the implantation due to the fact that recipient hepatectomy usually takes 2 hours. During this procedure, hypothermic oxygenated perfusion (HOPE group) for one hour will be performed vs continued cold storage (Control group).

We will use commercially available and approved IGL solution (Institut George Lopez) as perfusate for machine perfusion.

Subjects will be followed for one year after transplantation.

10 European centers are participating in this study, Randomization is stratified by center.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients with acute liver failure or liver cirrhosis (CHILD A, B or C) and/ or malignant liver tumors requiring liver transplantation
* Whole liver graft
* Signed informed consent

Exclusion Criteria:

* Split graft
* Living donor liver transplantation
* Grafts donated after cardiac arrest (DCD grafts)
* Domino transplantation
* Combined liver transplant
* Cold storage > 15h
* acute and unexpected medical contraindication

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-04; Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
major complications after liver transplantation | During the first year postoperatively
  post transplant complication Clavien >= III within 1 year after transplant

SECONDARY OUTCOMES:
Laboratory parameters post transplant | during first week, & 3,6,9,12 months
  Serum concentrations of bilirubin, AST, ALT, INR; Factor V
Cholangiopathy | during 12 months after transplant
  Biliary complications
hospital stay, ICU stay | during 12 months after transplant
  length of hospital and ICU stay after liver transplantation
Patient and graft survival | during 12 months after transplant
  one year patient and graft survival

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Dutkowski, Principal Investigator — Department of Surgery and Transplantation, University Hospital Zurich
Locations (2):
- Switzerland (2):
  - University Hospital of Zurich, Zurich
  - University of Zurich, Zurich

REFERENCES:
- [Background] de Rougemont O, Breitenstein S, Leskosek B, Weber A, Graf R, Clavien PA, Dutkowski P. One hour hypothermic oxygenated perfusion (HOPE) protects nonviable liver allografts donated after cardiac death. Ann Surg. 2009 Nov;250(5):674-83. doi: 10.1097/SLA.0b013e3181bcb1ee. PMID 19806056
- [Background] Dutkowski P, de Rougemont O, Clavien PA. Machine perfusion for 'marginal' liver grafts. Am J Transplant. 2008 May;8(5):917-24. doi: 10.1111/j.1600-6143.2008.02165.x. PMID 18416733
- [Background] Dutkowski P, Furrer K, Tian Y, Graf R, Clavien PA. Novel short-term hypothermic oxygenated perfusion (HOPE) system prevents injury in rat liver graft from non-heart beating donor. Ann Surg. 2006 Dec;244(6):968-76; discussion 976-7. doi: 10.1097/01.sla.0000247056.85590.6b. PMID 17122622
- [Derived] Schlegel A, Mueller M, Muller X, Eden J, Panconesi R, von Felten S, Steigmiller K, Sousa Da Silva RX, de Rougemont O, Mabrut JY, Lesurtel M, Cerisuelo MC, Heaton ND, Allard MA, Adam R, Monbaliu D, Jochmans I, Haring MPD, Porte RJ, Parente A, Muiesan P, Kron P, Attia M, Kollmann D, Berlakovich G, Rogiers X, Petterson K, Kranich AL, Amberg S, Mullhaupt B, Clavien PA, Dutkowski P. A multicenter randomized-controlled trial of hypothermic oxygenated perfusion (HOPE) for human liver grafts before transplantation. J Hepatol. 2023 Apr;78(4):783-793. doi: 10.1016/j.jhep.2022.12.030. Epub 2023 Jan 19. PMID 36681160